CLINICAL TRIAL: NCT05837585
Title: The Effectiveness of Air Quality Sensor on Resident Wellbeing and Changes in Care Routines in Elderly Residential Setting: A Single Group Pre-post Test Study
Brief Title: The Effectiveness of Air Quality Sensor in Elderly Residential Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Smart environment_protocol_v1
Record Dates: First submitted 2023-03-16; First posted 2023-05-01 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Technology; Signs and Symptoms, Respiratory
Keywords: Gerontechnology; Air quality sensor; Air quality improvement
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: The air quality sensors will install at the designated places and only serve to provide air quality indexes for the study site to improve air quality. The sensors will detect air quality at 2 weeks during the pre-test period and the alarm threshold will be set base on the 2-week data. During the 12 weeks trial period, based on the analysis on past 2-week air quality indexes, the managers of service unit will decide the changes of activities to improve air quality and long-term measures. The respiratory symptoms, blood pressure, pulse rate of participants will be collected during the pre-test and trial period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air quality sensors (Experimental): The experimental group will use the air quality sensors during 2 weeks pre-test and 12 weeks trial period.
  Interventions: Device: Air quality sensors

INTERVENTIONS:
Device: Air quality sensors — The air quality sensors detect air quality, including temperature, humidity, carbon dioxide, respirable suspended particulates (PM10 or PM2.5), total volatile organic compounds (TVOC) and formaldehyde (HCHO), which may influence health of residences. The managers of the service unit will decide the changes of activities to improve air quality and long-term measures based on the detected air quality indexes. The care staff will follow these decisions.

SUMMARY:
The study has 7 research questions regarding the use of the air quality sensor in residential care home for the elderly:

Primary study questions:

1. Can the real-time monitoring of air quality and the subsequent activities to improve air quality and long-term measures reduce respiratory symptoms?

   Secondary study questions:
2. Can the real-time monitoring of air quality and the subsequent activities to improve air quality and long-term measures reduce pulse rate, systolic blood pressure and diastolic blood pressure?
3. What are the activities to improve air quality and long-term measures that aim to improve air quality, including the rationales for change and non-change of the measures?
4. What are the changes in air quality indexes recorded by the air quality sensor?

   Auxiliary study questions:
5. How many days do the residents feel sick and stay in hospitals?
6. What are the perceived benefits and feasibility of the air quality sensor?

DETAILED DESCRIPTION:
Study design

The trial is a single group pre-post test study at Haven of Hope Woo Ping Care and Attention Home. There will be a pre-test of 2 weeks and trial of 12 weeks. During pre-test, the service unit will use the sensors to detect air quality. During the trial period, based on the analysis on air quality indexes in the past 2 weeks, the managers of the service unit will decide the changes of activities to improve air quality (e.g. opening windows, switching on fresh air supply fans and air purifiers, etc.) and long-term measures (e.g. using materials or plants that improve air quality, rearrange the bedroom, reschedule use of the rooms and activity schedule, replace air purifiers filters regularly, etc.) that may improve air quality.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Procedures

1. System installation

   The supplier will first visit the service unit(s) to determine the areas that probably have the worst air quality (usually these places are where many people gather yet lack ventilation). After confirming with the service unit managers, the sensors will be installed at the designated places. Related software(s) will be installed in computers in the nurse stations. The service unit(s) and the product supplier shall discuss the installation plan.
2. Participants' selection and consent

   The care staff will screen the appropriate residents with the eligibility criteria. The care staff will notify the eligible residents face-to-face individually about the air quality sensor and study. Their next of kin will be informed of the new devices and the study through standard channel of the test site (i.e. messaging mobile phone app or phone). If they do not want the residents to participate, they can notify the care staff. Unless they indicate withdrawal from the study, they are treated as consenting the residents to join the study (opt-out participation). The participants and their next of kins could request removal of the sensors and withdraw from the study at any time.

   Opt-out is considered sufficient to protect the rights of the vulnerable subjects. The air quality sensors only serve to provide additional information for the study site to improve care delivery. All measures taken to improve the air quality are determined by the study sites and not by the research. The participants and their next of kin can express their objections to the measures directly to the staff. The comments handling procedures adopted in daily care will be followed, such that when the study site sees it the best interest of the residents, the measures will be modified or terminated. The sensors will be installed in locations out of touch by the residents. They are light grey in colour and will not capture their attention.

   Before qualitative interviews with the participants and the staff, written consent will be obtained from them.
3. Pre-test

   The service unit will use the sensors to detect air quality for the first 2 weeks. The data will be reviewed to see if the readings are plausible. At the end of the pre-test, the staff will record the frequency of respiratory symptoms, including coughing, having sputum, having shortness of breath, and having runny nose, of the participants. Blood pressure and pulse rate are collected as a care routine of the test site and retrieved as secondary data. The research team, the supplier and the manager of the test site will analyze and review the air quality during the pre-test. An alarm threshold will be set for the 12-week trial period.
4. Implementation and data collection

During the pre-test and 12-week trial period, if the alert thresholds are set, when the air quality index is worse than the threshold, an alert will go off, and the staff will try to find out and document the possible reasons for worsened air quality. The care staff will take appropriate actions to improve air quality (e.g. moving the materials that are suspected to worsen air quality, report to the managers of service unit(s)). For the participants with respiratory and pulmonary illnesses, at the end of week 2, week 4, week 6, week 8, week 10 and week 12, the staff will record their respiratory symptoms. For other participants, their respiratory symptoms will be recorded at the end of week 2, week 4, week 8 and week 12. The University of Hong Kong (HKU) will assist analyzing the air quality of past 2 weeks retrieved from the air quality sensor. Based on the analysis, with the aim of improving air quality, the managers of the service unit(s) will decide the changes of activities to improve air quality (e.g. opening windows, switching on fresh air supply fans and air purifiers, etc.) and long-term measures (e.g. using materials or plants that improve air quality, rearrange the bedroom, reschedule use of the rooms and activity schedule, etc.) in the next 2 weeks. These changes, including the rationales for change and non-change in the measures, will be documented in decision records.

The number of sick days and hospital days of the residents in the previous 12 weeks will be retrieved at the end of the pre-test and 12-week trial.

At the end of the trial, qualitative interviews will be conducted to assess the perceived benefits and feasibility of the air quality sensor. A total of 2 to 3 residents and 2 to 5 staff will be interviewed.

Blinding

No blinding will be done for this single group study.

Sample size determination

The sample size is estimated by the number of air quality sensors and the number of residents staying in rooms with these sensors installed. It is expected that 60 elderly persons will join the study, and 2 - 5 care staff will be interviewed.

Data analyses

1. Main analysis

   Linear mixed modeling will be used to examine the changes in respiratory symptoms, pulse rate, systolic blood pressure, diastolic blood pressure, and the air quality indexes. Independent sample t-test will be used to test the difference of the number of sick days and hospital days of participants between pre-test and 12-week trial period.
2. Process evaluations

   The activities of air quality improvement and long-term measures decided by the managers of the service unit(s) will be summarized.
3. Qualitative interview

The interview content will be transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will be analyzed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the smart environment monitoring system. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of residents:

* Reside on the floor of the study site that will be installed with the air quality sensors, and
* Preferably have respiratory and pulmonary illnesses

Inclusion criteria of care staff:

* Responsible for the general care of the participants

Exclusion Criteria:

Exclusion criteria of residents and care staff:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline respiratory symptoms every two weeks until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  Change of four respiratory symptoms of participants, including coughing, having sputum, having shortness of breath and having runny nose, will be observed and recorded by the care staff every two weeks. Care staff will complete four items on a 5-point Likert scale (i.e. 1 indicating no symptoms and 5 indicating serve symptoms). The minimum and maximum values of the scale is 5 and 25 respectively, with higher score indicating more severe respiratory symptoms.

SECONDARY OUTCOMES:
Change from Baseline pulse rate every week until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  Change of pulse rate in beats per minute (bpm) of participants will be collected as a care routine of the service unit(s) every week and retrieved as secondary data.
Change from Baseline blood pressure every week until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  Change of systolic blood pressure and diastolic blood pressure in millimeters of mercury (mmHg) of participants will be collected as a care routine of the service unit(s) every week and retrieved as secondary data.
Qualitative measures: Change of air quality improvement measures every two weeks until week 14 | From the end of 2-week pre-test to the end of 12-week trial period
  Qualitative change of air quality improvement measures (e.g. using materials or plants, relocating the air purifiers, reschedule use of the rooms, etc.) will be decided and documented in decision records by the managers of service unit(s) every two weeks. The list of air quality improvement measures is not exhaustive and managers could be creative in designing the measures.
The changes in temperature until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The temperature in degrees Celsius (℃) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in humidity until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The humidity in percentage (%) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in carbon dioxide until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The carbon dioxide in parts per million (ppm) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in respirable suspended particulates (PM2.5) until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The respirable suspended particulates (PM2.5) in micrograms per cubic meter (µg/m3) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in total volatile organic compounds (TVOC) until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The total volatile organic compounds (TVOC) in part per billion (ppb) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in formaldehyde until week 14 | From the start of 2-week pre-test to the end of 12-week trial period
  The formaldehyde in part per billion (ppb) of testing areas will be recorded by the sensor system continuously until week 14.
The changes in the number of sick days of participants between 12 weeks before the trial and trial period | From 12 weeks before the trial to the end of 12-week trial period
  The number of sick days of the participants in 12 weeks before the trial and trial period will be retrieved from residency reports.
The number of hospital days of participants between 12 weeks before the trial and trial period | From 12 weeks before the trial to the end of 12-week trial period
  The number of hospital days of participants in 12 weeks before the trial and trial period will be retrieved from residency reports.
Qualitative measures: The perceived benefits and feasibility of the air quality sensor of residents | At the end of 12-week trial period
  Qualitative interviews will be conducted to assess the perceived benefits and feasibility of the air quality sensor. 2 to 3 residents will be interviewed and the contents including:
  1. Do you think the air quality sensor is safe?
  2. Is there any changes of your respiratory symptoms?
  3. Do you feel any inconvenience during the changes of activities to improve air quality?
  4. Are you satisfied with the air quality sensor?
  5. Do you want the service unit to continue to use air quality sensor?
Qualitative measures: The perceived benefits and feasibility of the air quality sensor of care staff | At the end of 12-week trial period
  Qualitative interviews will be conducted to assess the perceived benefits and feasibility of the air quality sensor. 2 to 5 care staffs will be interviewed and the contents including:
  1. Do you think the air quality sensor is safe?
  2. Is it difficult to understand the air quality report?
  3. Does the air quality sensor affect your daily routine?
  4. Did the air quality sensor detect the change in air quality after the activities to improve air quality were implemented?
  5. Do you think the air quality indexes can be used to define air quality in the environment?
  6. Are there other benefits of the air quality sensor besides the real-time monitoring on air quality?
  7. Do you think it is easy to find out the causes of the worsened air quality with reference to the air quality indexes?
  8. What are the burden while implementing the activities to improve air quality?
  9. On the whole, are you satisfied with the sensors?
  10. To what extent, do you want to continue to use the sensors?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Haven of Hope Woo Ping Care & Attention Home, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.